CLINICAL TRIAL: NCT04776694
Title: Compassionate Use of Dupilumab
Status: Approved for marketing | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-Dupilumab
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Inflammatory Disorders
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Dupilumab
  Other Names: REGN668; DUPIXENT®; SAR231893

SUMMARY:
Provide Compassionate Use of Dupilumab

DETAILED DESCRIPTION:
Compassionate Use requests are only being considered in response to Individual Patient Investigational New Drug (IND) applications. Availability will depend on location.

Age Groups: Child, Adult, Older Adult